CLINICAL TRIAL: NCT02903628
Title: Vice-president, Nurse, Principal Investigator
Brief Title: The Model Building and Empirical Research of Eye Health Interventions for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Chen yanyan, Vice-president, Nurse, Principal Investigator, Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2012C3301
Record Dates: First submitted 2016-09-04; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Myopia
Keywords: myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- eye health education (Experimental)
  Interventions: Behavioral: eye health education

INTERVENTIONS:
Behavioral: eye health education — give a lecture and issue knowledge manual for children and parents ,6 months once , 2.5 years

SUMMARY:
The purpose of this study is to determine whether Eye Health Intervention can obviously reduce and delay myopia onset and development and improved the awareness rate of knowledge apparently .

ELIGIBILITY:
Inclusion Criteria:

* primary 1-3 grade students

Exclusion Criteria:

* ocular inflammation
* eye injury
* dysgnosia

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1517 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of Myopia | every 6 months, total 3 years

SECONDARY OUTCOMES:
health of eyes knowledge | every 6 months, total 3 years, questionnair
health of eyes behavior | every 6 months, total 3 years, questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: yan yan chen, master, Study Chair — Wenzhou Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Leo SW, Young TL. An evidence-based update on myopia and interventions to retard its progression. J AAPOS. 2011 Apr;15(2):181-9. doi: 10.1016/j.jaapos.2010.09.020. PMID 21596297
- [Result] Saw SM, Shih-Yen EC, Koh A, Tan D. Interventions to retard myopia progression in children: an evidence-based update. Ophthalmology. 2002 Mar;109(3):415-21; discussion 422-4; quiz 425-6, 443. doi: 10.1016/s0161-6420(01)00972-1. PMID 11874738
- [Result] Schaeffel F. [Myopia update 2011]. Klin Monbl Augenheilkd. 2011 Sep;228(9):754-61. doi: 10.1055/s-0031-1281584. Epub 2011 Jul 27. German. PMID 21796575
- [Result] Adler D, Millodot M. The possible effect of undercorrection on myopic progression in children. Clin Exp Optom. 2006 Sep;89(5):315-21. doi: 10.1111/j.1444-0938.2006.00055.x. PMID 16907670
- [Result] Seet B, Wong TY, Tan DT, Saw SM, Balakrishnan V, Lee LK, Lim AS. Myopia in Singapore: taking a public health approach. Br J Ophthalmol. 2001 May;85(5):521-6. doi: 10.1136/bjo.85.5.521. No abstract available. PMID 11316705